CLINICAL TRIAL: NCT04582890
Title: US Time-Harmonic Elastography for the Early Detection of Childhood Glomerulonephritis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Mostafa Sayed Mostafa, Resident doctor, Assiut University
Other Study IDs: Glomerulonephritis
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
US Time-Harmonic Elastography for the Early Detection of Childhood Glomerulonephritis

DETAILED DESCRIPTION:
Glomerulonephritis (GN) comprises a group of renal diseases characterized by glomerular and tubulointerstitial fibrosis secondary to glomerular inflammation and proliferation of the basement membrane, mesangial cells, or capillary endothelium triggered by immunologic mechanisms.(1) The glomerular filtration rate decreases with progression of chronic kidney disease (CKD), ultimately resulting in end-stage renal failure. Glomerulonephritis is the third most common cause of end-stage renal failure. Initial clinical signs of glomerulonephritis are nonspecific and subtle. Occasionally, affected patients present with hypertension, proteinuria, hematuria, raised serum creatinine level, weight gain, edema, or nephrotic syndrome.(2) The underlying pathologic changes are partly irreversible, and a prompt diagnosis with early initiation of treatment is of vital importance. The diagnosis is based on clinical, laboratory, and conventional US findings, whereas renal biopsy is considered the reference standard for a definitive diagnosis and fibrosis grading.(3,4) Unfortunately, this invasive procedure is associated with the risk of serious bleeding complications and therefore is not the method of choice for longitudinal monitoring.

Elastography, a Novel imaging modality that estimates tissue stiffness, especially for superficial organs such as the breast and Thyroid. In recent years, ultrasound elastography (UE) has been demonstrated in the liver and has been applied widely in the diagnosis and evaluation of liver diseases, such as chronic hepatitis, alcoholic liver diseases, and non alcoholic fatty liver diseases.(5,6) To date, renal allograft stiffness (elasticity) has been evaluated by magnetic resonance elastography (MRE) and ultrasound elastography (UE). However, UE application for native renal diseases has not been well up till now.(7) Conventional renal ultrasonography may be appropriate to evaluate kidney size, as well as to assess the echogenicity of the renal cortex, exclude obstruction, and determine the extent of fibrosis. However, It has no significant role in diagnosis of GN. US time-harmonic elastography depicts abnormal renal stiffness in glomerulonephritis, particularly among patients with early disease and preserved renal function.(8,9,10)

ELIGIBILITY:
Inclusion Criteria:

1. Age 1 month up to 18 years
2. Patientswith acute glomerulonephritis either poststreptococcal , lupus, ANCA related, or Ig A nephritis . Diagnosis of such diseases will be done through usual clinical, laboratory , radiological and histopathological data

Exclusion Criteria:

patients with clinical, laboratory , or radiological evidence of chronic kidney disease

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patientswith acute glomerulonephritis either poststreptococcal , lupus, ANCA related, or Ig A nephritis . Diagnosis of such diseases will be done through usual clinical, laboratory , radiological and histopathological data
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
The diagnostic performance of US time-harmonic elastography for the early detection of glomerulonephritis will be assessed with calculation of its sensitivity ,specificity and accuracy | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol